CLINICAL TRIAL: NCT02012231
Title: A Phase I/IIa Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of PLX8394 in Patients With Advanced, Unresectable Solid Tumors
Brief Title: Phase I/IIa Study to Evaluate the Safety, PK, PD, and Preliminary Efficacy of PLX8394 in Patients With Advanced Cancers.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Fore Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLX120-01
Record Dates: First submitted 2013-12-05; First posted 2013-12-16 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2016-05

CONDITIONS: Melanoma; Thyroid Cancer; Colorectal Cancer; Non-small Cell Lung Cancer; Cholangiocarcinoma; Histiocytosis; Hairy Cell Leukemia
Keywords: melanoma; anaplastic thyroid cancer; advanced papillary thyroid cancer; colorectal cancer; non-small cell lung cancer; cholangiocarcinoma; histiocytosis; hairy cell leukemia
MeSH Terms: conditions — Melanoma; Thyroid Neoplasms; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Cholangiocarcinoma; Histiocytosis; Leukemia, Hairy Cell; Thyroid Carcinoma, Anaplastic | interventions — PLX8394

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose Escalation (Experimental): Cohort 1/Day -7 = 300 mg/day PLX8394; Cohort 1/Day 1 = 900 mg/day PLX8394
  Interventions: Drug: PLX8394

INTERVENTIONS:
Drug: PLX8394 — PLX8394 is a next-generation, orally available, small-molecule, selective inhibitor of BRAF.

SUMMARY:
The study objective is to evaluate the safety, pharmacokinetics (PK), and pharmacodynamics (PD) of orally administered PLX8394 in patients with advanced solid tumors. An additional objective is to identify a Recommended Phase 2 (RP2D) for further evaluation in the Extension Cohorts (Phase IIa portion).

The study objective of the Extension Cohorts (PART 2 portion) is to assess the objective tumor response and the PK, PD, and safety of PLX8394 when the RP2D is used in patients with advanced BRAF-mutated cancers.

DETAILED DESCRIPTION:
This is an open-label, multi-center Phase I/IIa two-part study with a sequential dose escalation part, followed by three parallel Extension cohorts (BRAF-mutated melanoma, BRAF-mutated non-melanoma solid tumors, and BRAF-mutated classical hairy cell leukemia). Up to approximately 42 patients may be enrolled in the dose escalation phase of the study, depending on the number of cohorts required, number of patients per cohort needed, and the need for replacement patients. Approximately 130 patients are planned to be enrolled in the BRAF-mutated tumor Extension cohorts, with the goal of enrolling approximately 50 patients with BRAF/MEK/ERK inhibitor-naïve melanoma, approximately 10-15 patients with BRAF/MEK/ERK inhibitor-pretreated melanoma, approximately 50 patients with non-melanoma solid tumors, and approximately 10-15 patients with hairy cell leukemia. The trial was intended to be a Phase 1/2 trial, but the trial never moved forward to Phase 2.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Measurable disease by RECIST 1.1 criteria (solid tumors)
* ECOG performance status of 0-2
* Life expectancy ≥ 3 months
* Adequate hematologic, hepatic, and renal function:

  1. Solid Tumors - Absolute neutrophil count ≥ 1.5 × 109/L, Hgb > 9 g/dL, platelet count ≥ 100 × 109/L, AST/ALT ≤ 2.5 × ULN, bilirubin ≤ 2, creatinine ≤ 1.5 × ULN or calculated CrCl >50 mL/min (Cockcroft-Gault formula)
  2. Hairy Cell Leukemia - Absolute neutrophil count ≤ 1.0 × 109/L, Hgb ≤ 10.0 g/dL or platelet count ≤ 100 × 109/L; AST/ALT ≤ 2.5 × ULN, bilirubin ≤ 2, creatinine ≤ 1.5 × ULN or calculated CrCl >50 mL/min (Cockcroft-Gault formula)
* Women of child-bearing potential must have a negative serum pregnancy test within 14 days of initiating study drug and must agree to use an acceptable method of birth control from the time of the negative pregnancy test up to 6 months after the last dose of study drug. Urine pregnancy testing during the study and in follow-up per country specific requirements. Fertile men must also agree to use an acceptable method of birth control while on study drug and up to 6 months after the last dose of study drug.
* Completion of previous chemotherapy, immunotherapy, or radiation therapy at least 2 weeks before study drug initiation, with resolution of all associated toxicity (to ≤ Grade 1 or Baseline)
* Willingness and ability to provide written informed consent prior to any study-related procedures and to comply with all study requirements
* Eligibility for medical insurance coverage

  1. DOSE-ESCALATION COHORTS
* advanced solid tumors that are refractory to standard therapy, have no standard therapy, or are considered by the investigator to be inappropriate for standard therapy

  2. EXTENSION COHORTS
* Cancers with a BRAF-activating mutation as assessed by a CLIA-certified method

  a. Melanoma
* unresectable Stage IIIC or Stage IV disease (sub-cohort 1a: BRAF/MEK/ERK inhibitor naïve, sub-cohort 1b: BRAF/MEK/ERK inhibitor pre-treated) b. Non-melanoma Solid Tumors
* advanced anaplastic thyroid cancer, advanced papillary thyroid cancer, and advanced solid tumors (e.g., colorectal cancer, non-small cell lung cancer, cholangiocarcinoma, etc) that are refractory to standard therapy, relapsed after standard therapy, have no standard therapy, or are considered by the investigator to be inappropriate for standard therapy c. Hairy Cell Leukemia
* histologically confirmed classical hairy cell leukemia that failed to achieve CR or PR to initial purine analog-based therapy, relapsed ≤ 2 years after purine analog-based therapy, or a history of intolerance to purine analogs

Exclusion Criteria:

* Extension Cohorts (except 1b) - Previous treatment with a selective BRAF/MEK/EKR inhibitor
* Symptomatic brain metastases. Patients with untreated brain metastasis ≤ 1 cm can be considered eligible if deemed asymptomatic by the investigator upon consultation with the medical monitor and do not require immediate radiation or steroids. Patients with brain metastasis that is treated and stable for 1 month may be considered eligible if they are asymptomatic and on stable dose of steroids or if they do not require steroids following successful local therapy.
* Investigational drug use within 28 days (or < 5 half-lives, whichever is shorter) of the first dose of PLX8394
* Major surgical procedure, open biopsy (excluding skin cancer resection), or significant traumatic injury within 14 days of initiating study drug (unless the wound has healed) or anticipation of the need for major surgery during the study
* Uncontrolled intercurrent illness
* Active secondary malignancy unless the malignancy is not expected to interfere with the evaluation of safety and is approved by the Medical Monitor. Examples of the latter include basal or squamous cell carcinoma of the skin, in-situ carcinoma of the cervix, and isolated elevation of prostate-specific antigen. Patients with a completely treated prior malignancy and no evidence of disease for ≥ 2 years are eligible.
* Refractory nausea and vomiting, malabsorption, external biliary shunt, or significant bowel resection that would preclude adequate absorption
* Baseline mean QTcF ≥ 450 ms (males) or ≥ 470 ms (females)
* Women who are breast-feeding or pregnant
* Known chronic HIV, HCV, or HBV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Phase 1 dose escalation: Identification of Recommended Phase 2 Dose Safety of PLX8394 | 1 Year
  Physical examinations, vital signs, 12-lead electrocardiograms, adverse events, hematology, serum chemistry, and urinalysis will be used to assess safety and tolerability.

SECONDARY OUTCOMES:
Identification of Recommended Phase 2 dose (RP2D) | 1 year
  Study drug administration is dosed continuously until clinically significant disease progression, discontinuation of study for any reason or one of the stopping criteria is met.

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Sharma, MD, Principal Investigator — Huntsman Cancer Institute
Locations (3):
- United States (3):
  - Scottsdale Healthcare, Scottsdale, Arizona
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Evergreen Hematology & Oncology, Spokane, Washington